CLINICAL TRIAL: NCT06969222
Title: A Prospective Clinical Investigation of Robotic-assisted TKA (RA-TKA) With Skywalker and Evolution Medial Pivot Knee (eMP Knee)
Brief Title: l Investigation of Robotic-assisted TKA (RA-TKA) With Skywalker and Evolution Medial Pivot Knee (eMP Knee)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Department of General University Hospital of Laria (Other)
Collaborators: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Principal Investigator, Theofilos Karachalios, Professor of Orthopaedics, Head of Orthopaedic Department, University Hospital of Larisa, Orthopaedic Department of General University Hospital of Laria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 50377/24-11-22
Record Dates: First submitted 2023-10-02; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Knee Arthropathy; Arthroplasty Complications; Robotic Assisted Arthroplasty; TKA Outcomes
Keywords: knee arthroplasty; Skywalker robotic System; evolution medial pivot implant

STUDY DESIGN:
Intervention Model Description: prospective randomized trial with 122 patients divided into two groups One operated with robotic-assisted arthroplasty and other operated with conventional total knee arthroplasty
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic-assisted Skywalker device - Evolution Medial Pivot (Active Comparator)
  Interventions: Procedure: Robotic TKA
- Conventional total knee arthroplasty with manual instruments - device - Evolution Medial Pivot (Active Comparator)

INTERVENTIONS:
Procedure: Robotic TKA — Total knee replacement of arthritic knees either with robotic-assisted Skywalker device
  Arms: Robotic-assisted Skywalker device - Evolution Medial Pivot
Procedure: Conventional TKA — Total knee replacement of arthritic knees performed manually

SUMMARY:
This is a prospective trial that attempts to develop evidence on the safety and performance of RA-TKA (Robotic-assisted total knee arthroplasty) with Skywalker and eMP (Evolution Medial Pivot) knee. Moreover to evaluate performance of eMP patients with Skywalker (in comparison to eMP with conventional instrumentations and non-MP TKAs)

DETAILED DESCRIPTION:
The included patients will be those who meet study inclusion and exclusion criteria (IEC) to receive RA-TKA with Skywalker and eMP knees. This cohort will include learning curve cases from each surgeon. The learning curve cases will be determined based on the assessment of parameters such as surgical time etc.

Patients who have received eMP knees with conventional instrumentations or non-MP TKAs (retrospective)

Inclusion Criteria:

1. >= 18 Years Male or Female
2. With noninflammatory degenerative joint disease, inflammatory joint disease, functional deformity
3. The subject has signed the Ethical Board approved Informed Consent Form specific to this study prior to enrollment
4. Must be independent, ambulatory, and can comply with all post-operative evaluations and visits.

Exclusion Criteria:

1. Subjects with poor compliance, unable to complete the trial according to the requirements or for other reasons or considered not to be suitable for inclusion by investigators.
2. Concurrent participation in any other total hip or knee replacement studies.

Study Objectives: Evaluate Safety and Performance of RA-TKA with Skywalker and eMP knee and address research questions include but not limited to:

1. Accuracy and Reproducibility of Skywalker with eMP knee
2. Learning Curve of adopting Skywalker with eMP knees
3. Postop function recovery in eMP patients with Skywalker
4. Safety of eMP knee with Skywalker based on intra-op and postop complications
5. (Enhanced) Kinematics of eMP with Skywalker compared to manual and other non MP TKA

Study Endpoints Primary Effectiveness Endpoints

* FJS and OKS at 12 months
* Kinematics from RSA at min 6 months

Primary Safety Endpoint

* Revisions / surgical interventions including MUA on the index knee due to any reasons
* Serious Adverse Events that require hospitalization

Secondary Endpoint

* Accuracy based on planned vs actual size and alignment parameters
* FJS at 6 weeks, 3 months, 6 months
* OKS at 6 weeks, 3 months, 6 months
* ROM from KSS at 6 weeks, 6 months and 12 months
* Learning Curve based on surgical time

ELIGIBILITY:
Inclusion Criteria:

1. >= 18 Years Male or Female
2. With noninflammatory degenerative joint disease, inflammatory joint disease, functional deformity
3. The subject has signed the Ethical Board approved Informed Consent Form specific to this study prior to enrollment
4. Must be independent, ambulatory, and can comply with all post-operative evaluations and visits.

Exclusion Criteria:

1. Subjects with poor compliance, unable to complete the trial according to the requirements or for other reasons or considered not to be suitable for inclusion by investigators.
2. Concurrent participation in any other total hip or knee replacement studies.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 122 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoints with outcome scores Primary Effectiveness Endpoints | 2 years after intervention
  KOOS score(Knee Injury and Osteoarthritis Outcome Score) with a 0-100 scale measured at 1, 3, 6 and 12 months
Primary Effectiveness Endpoints with outcome scores Primary Effectiveness Endpoints | 2 years after intervention
  FJS (Forgotten Joint Score) with a scale 0 to 48 score measured at 1, 3, 6, and 12 months
Primary Effectiveness Endpoints with outcome scores Primary Effectiveness Endpoints | 2 years after intervention
  VAS score (Visual Analogue Scale) with a 0-10 scale measured at 1, 3, 6 and 12 months
Primary Effectiveness Endpoints with outcome scores Primary Effectiveness Endpoints | 2 years after intervention
  OKS score(Oxford Knee Score) with a 0-100 scale measured at 1, 3, 6 and 12 months
Primary safety endpoints | 1 year after intervention
  Revisions / surgical interventions including MUA on the index knee due to any reason. Severe adverse effects

SECONDARY OUTCOMES:
Accuracy of implantation measured in degrees of correction | 1 year after intervention
  Accuracy based on planned vs actual size and alignment parameters
Learning curve | 1 year after intervention
  Learning curve based on surgical time

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Larisa, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karachalios T, Varitimidis S, Bargiotas K, Hantes M, Roidis N, Malizos KN. An 11- to 15-year clinical outcome study of the Advance Medial Pivot total knee arthroplasty: pivot knee arthroplasty. Bone Joint J. 2016 Aug;98-B(8):1050-5. doi: 10.1302/0301-620X.98B8.36208. PMID 27482016
- [Background] St Mart JP, Goh EL. The current state of robotics in total knee arthroplasty. EFORT Open Rev. 2021 Apr 1;6(4):270-279. doi: 10.1302/2058-5241.6.200052. eCollection 2021 Apr. PMID 34040804
- [Background] Siddiqi A, Horan T, Molloy RM, Bloomfield MR, Patel PD, Piuzzi NS. A clinical review of robotic navigation in total knee arthroplasty: historical systems to modern design. EFORT Open Rev. 2021 Apr 1;6(4):252-269. doi: 10.1302/2058-5241.6.200071. eCollection 2021 Apr. PMID 34040803